CLINICAL TRIAL: NCT05414266
Title: A Randomized, Placebo Controlled Single Site Study Evaluating Efficacy of Topical Squaric Acid Dibutyl Ester in Children and Adolescents With Alopecia Areata
Brief Title: Study Evaluating Efficacy of Topical Squaric Acid Dibutyl Ester in Children and Adolescents With Alopecia Areata
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Adelaide Hebert, Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HSC-MS-21-1035
Record Dates: First submitted 2022-06-07; First posted 2022-06-10 (Actual); Last update posted 2022-10-13 (Actual); Status verified 2022-10

CONDITIONS: Alopecia Areata
Keywords: Alopecia
MeSH Terms: conditions — Alopecia Areata; Alopecia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 4 months Placebo, then 8 months SADBE 5% (Experimental)
  Interventions: Drug: Placebo; Drug: SADBE 5%
- 12 months SADBE 5% (Experimental)
  Interventions: Drug: SADBE 5%

INTERVENTIONS:
Drug: Placebo — Placebo is acetone. At baseline, the investigator will record the area that will be treated in mm2 . Use of a 1 mm x 1 mm gridded transparency will be used to record the treatment area at baseline. At subsequent visits, the study intervention will be applied to the entire treatment area defined at baseline, regardless of any new hair growth. The assigned study intervention is applied monthly by the PI (or designee) to the treatment areas affected by AA on the scalp and/or eyebrows identified at Baseline. The topical solution is applied with a cotton tip applicator by the PI or their qualified designee. Solution is applied by gently pressing a cotton tip applicator that has been soaked in the study solution against the skin. Treatment is repeated monthly.
  Arms: 4 months Placebo, then 8 months SADBE 5%
Drug: SADBE 5% — SADBE 5% is a solution of 5% Squaric Acid Dibutyl Ester (SADBE) in acetone. At baseline, the investigator will record the area that will be treated in mm2 . Use of a 1 mm x 1 mm gridded transparency will be used to record the treatment area at baseline. At subsequent visits, the study intervention will be applied to the entire treatment area defined at baseline, regardless of any new hair growth. The assigned study intervention is applied monthly by the PI (or designee) to the treatment areas affected by AA on the scalp and/or eyebrows identified at Baseline. The topical solution is applied with a cotton tip applicator by the PI or their qualified designee. Solution is applied by gently pressing a cotton tip applicator that has been soaked in the study solution against the skin. Treatment is repeated monthly.

SUMMARY:
The purpose of this study is to evaluate the efficacy and tolerability of squaric acid dibutylester (SADBE) in children and adolescents with alopecia areata (AA) and to evaluate effect of squaric acid dibutyl ester on patient-centered outcomes and payer relevant measures to assess treatment benefit from the patient perspective and to demonstrate value

ELIGIBILITY:
Inclusion Criteria:

* Evidence of a personally signed and dated informed consent document indicating that the participant or a legally acceptable representative/parent(s)/legal guardian has been informed of all pertinent aspects of the study.
* Willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures.
* not pregnant or breast feeding
* Participants who are women of child bearing potential(WOCBP) must agree to use one highly effective method of contraception(with a failure rate of <1% per year during the intervention period and for at least 28 days after the last dose of study intervention.
* Negative highly sensitive pregnancy (urine) at the Day 1 visit before the first dose of study intervention for WOCBP
* Have a clinical diagnosis of AA with no other etiology of hair loss (e.g., telogen effluvium,androgenetic alopecia, etc.)
* greater than 10% hair loss of the scalp, including without evidence of terminal hair regrowth within 6 months at both screening and baseline visits
* Current episode of hair loss less than 5 years.
* must be on a stable regimen of permitted concomitant medication
* Must agree to avoid prolonged exposure to the sun and not to use tanning booths, sun lamps or other ultraviolet light sources in the treatment area during the study.

Exclusion Criteria:

* Other scalp disease that may impact AA assessment (e.g., scalp psoriasis, dermatitis, etc).
* Active systemic diseases that may cause hair loss (e.g., lupus erythematosus, thyroiditis, systemic sclerosis, lichen planus, etc).
* Any psychiatric condition including recent or active suicidal ideation or behavior
* Ongoing or recent history of any other uncontrolled and/or clinically significant medical or psychiatric disease or condition which, in the PI's medical opinion, should exclude participation in the study.
* Any present malignancies or history of malignancies with the exception of adequately treated or excised non metastatic basal cell or squamous cell cancer of the skin or cervical carcinoma in situ.
* History (single episode) of disseminated herpes zoster or disseminated herpes simplex, or a recurrent (more than one episode of) localized, dermatomal herpes zoster
* History of systemic infection requiring hospitalization, parenteral antimicrobial therapy, or as otherwise judged clinically significant by the investigator within 6 months prior to Day 1
* Known primary or secondary immunodeficiency disorder or a first-degree relative with a hereditary immunodeficiency
* Significant trauma or major surgery within 1 month of the first dose of study intervention.
* Considered in imminent need for surgery. Participants with elective surgery scheduled can only be enrolled in Study SADBE-high dose (HD) with the approval of the investigator.
* Active acute or chronic infection requiring treatment with oral antibiotics, antivirals, anti-parasitics, anti-protozoals, or antifungals within 4 weeks prior to Day 1 or any active systemic or local infection not meeting other exclusion criteria within 1 week prior to Day 1.
* Participant has a known hypersensitivity or previous allergic reaction to any of the active or inactive ingredients in the study intervention
* Anticipated treatment with prohibited concomitant medication(s) during the course of the study
* Received Herbal medications with either unknown properties or pharmaceutical properties that impact AA within 1 week of first dose of study intervention
* Received topical steroids (e.g., steroid cream, steroid ointment) on areas under assessment (i.e., scalp, eyebrows). within 2 week of first dose of study intervention
* Received Ultraviolet B (UVB) phototherapy, Psoralen Ultraviolet A (PUVA) therapy, other phototherapy, contact immunotherapy [e.g.diphenylcyclopropenone (DPCP), and 1-chloro-2,4-dinitrobenzene (DNCB)], topical irritants(e.g., anthralin), and liquid nitrogen cryotherapy within 4 weeks of first dose of study intervention
* Received Other topical or systemic treatments that could affect AA including: Immune suppressants (e.g., cyclosporine A, azathioprine, methotrexate (MTX), sulfasalazine, mycophenolate mofetil (MMF), everolimus, ibrutinib, Intralesional, topical, oral, or injectable (intramuscular or intraarticular)steroids or Oral or topical minoxidil within 8 weeks of first dose of study intervention or within 5 half-lives (if known), whichever is longer
* Received Any Janus kinase (JAK) inhibitor for use in any disease indication or other immunomodulatory biologic agents within 12 weeks of first dose of study intervention or 5 half-lives (if known), whichever is longer
* Investigator site staff members directly involved in the conduct of the study and their family members, site staff members otherwise supervised by the investigator, or participants who are University of Texas employees, including their family members, directly involved in the conduct of the study.
* Participants with shaved heads must not enter the study until hair has grown back to a reasonable level and is considered stable, in the opinion of the investigator.
* Have an active history of alcohol or substance abuse within 1 year prior to Day 1.
* Participant is unable to communicate or cooperate with the investigator due to language problems, poor mental development, or impaired cerebral function.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 36 (Estimated)
Dates: Start 2022-08-15 (Actual); Primary Completion 2023-06-01 (Estimated); Study Completion 2024-05-22 (Estimated)

PRIMARY OUTCOMES:
Hair loss as assessed by number of subjects that score <30 on the the Severity of alopecia tool (SALT) | end of treatment (12 months of treatment)
  The SALT measures the percentage of hair loss on the scalp utilizing a visual aid showing the division of the scalp hair into four quadrants (back, top of scalp, and both sides), with each of the four quadrants given an accurate determination of the % of scalp surface area covered, representing 24%, 40%, 18%, and 18% of the total scalp surface area, respectively.
  Total SALT score is reported and calculated as: Total SALT Score=[0.40x%scalp hair loss top quadrant]+[0.24x%scalp hair loss back quadrant]+[0.18x%scalp hair loss left quadrant]+[0.18x% scalp hair loss right quadrant]
Hair loss as assessed by the number of subjects that score <50 on the the Severity of alopecia tool (SALT) | month 4
  The SALT measures the percentage of hair loss on the scalp utilizing a visual aid showing the division of the scalp hair into four quadrants (back, top of scalp, and both sides), with each of the four quadrants given an accurate determination of the % of scalp surface area covered, representing 24%, 40%, 18%, and 18% of the total scalp surface area, respectively.
  Total SALT score is reported and calculated as: Total SALT Score=[0.40x%scalp hair loss top quadrant]+[0.24x%scalp hair loss back quadrant]+[0.18x%scalp hair loss left quadrant]+[0.18x% scalp hair loss right quadrant]
Overall hair loss as assessed by the SALT score | Baseline, Month 1, Month 2, Month 3, Month 4, Month 5, Month 6, Month 7, Month 8,Month 9, Month 10, Month 11, Month 12(end of treatment),Month 14(end of study),early termination visit (occurs only if subject discontinues form study)
  The SALT measures the percentage of hair loss on the scalp utilizing a visual aid showing the division of the scalp hair into four quadrants (back, top of scalp, and both sides), with each of the four quadrants given an accurate determination of the % of scalp surface area covered, representing 24%, 40%, 18%, and 18% of the total scalp surface area, respectively.
  Total SALT score is reported and calculated as: Total SALT Score=[0.40x%scalp hair loss top quadrant]+[0.24x%scalp hair loss back quadrant]+[0.18x%scalp hair loss left quadrant]+[0.18x% scalp hair loss right quadrant]
AA hair loss as assessed by the SALT score | Baseline, Month 1, Month 2, Month 3, Month 4, Month 5, Month 6, Month 7, Month 8,Month 9, Month 10, Month 11, Month 12(end of treatment),Month 14(end of study),early termination visit (occurs only if subject discontinues form study)
  The SALT measures the percentage of hair loss on the scalp utilizing a visual aid showing the division of the scalp hair into four quadrants (back, top of scalp, and both sides), with each of the four quadrants given an accurate determination of the % of scalp surface area covered, representing 24%, 40%, 18%, and 18% of the total scalp surface area, respectively.
  Total SALT score is reported and calculated as: Total SALT Score=[0.40x%scalp hair loss top quadrant]+[0.24x%scalp hair loss back quadrant]+[0.18x%scalp hair loss left quadrant]+[0.18x% scalp hair loss right quadrant]
Change in overall hair loss as assessed by the Severity of alopecia tool (SALT) | Baseline, Month 1,Month2,Month 3, Month 4, Month 5, Month 6, Month 7, Month 8,Month 9, Month 10, month 11, Month 12,Month 14,early termination visit (occurs only if subject discontinues form study)
  The SALT measures the percentage of hair loss on the scalp utilizing a visual aid showing the division of the scalp hair into four quadrants (back, top of scalp, and both sides), with each of the four quadrants given an accurate determination of the % of scalp surface area covered, representing 24%, 40%, 18%, and 18% of the total scalp surface area, respectively.
  Total SALT score is reported and calculated as: Total SALT Score=[0.40x%scalp hair loss top quadrant]+[0.24x%scalp hair loss back quadrant]+[0.18x%scalp hair loss left quadrant]+[0.18x% scalp hair loss right quadrant]
Change in AA hair loss as assessed by the Severity of alopecia tool (SALT) | Baseline, Month 1,Month2,Month 3, Month 4, Month 5, Month 6, Month 7, Month 8,Month 9, Month 10, month 11, Month 12,Month 14,early termination visit (occurs only if subject discontinues form study)
  The SALT measures the percentage of hair loss on the scalp utilizing a visual aid showing the division of the scalp hair into four quadrants (back, top of scalp, and both sides), with each of the four quadrants given an accurate determination of the % of scalp surface area covered, representing 24%, 40%, 18%, and 18% of the total scalp surface area, respectively.
  Total SALT score is reported and calculated as: Total SALT Score=[0.40x%scalp hair loss top quadrant]+[0.24x%scalp hair loss back quadrant]+[0.18x%scalp hair loss left quadrant]+[0.18x% scalp hair loss right quadrant]
Overall hair loss as assessed by the number of subjects with at least 50% improvement in the SALT score as assessed by the Severity of alopecia tool (SALT) | Baseline, Month 1, Month 2, Month 3, Month 4, Month 5, Month 6, Month 7, Month 8,Month 9, Month 10, Month 11, Month 12(end of treatment),Month 14(end of study),early termination visit (occurs only if subject discontinues form study)
  The SALT measures the percentage of hair loss on the scalp utilizing a visual aid showing the division of the scalp hair into four quadrants (back, top of scalp, and both sides), with each of the four quadrants given an accurate determination of the % of scalp surface area covered, representing 24%, 40%, 18%, and 18% of the total scalp surface area, respectively.
  Total SALT score is reported and calculated as: Total SALT Score=[0.40x%scalp hair loss top quadrant]+[0.24x%scalp hair loss back quadrant]+[0.18x%scalp hair loss left quadrant]+[0.18x% scalp hair loss right quadrant]
AA hair loss as assessed by the number of subjects with at least 50% improvement in the SALT score as assessed by the Severity of alopecia tool (SALT) | Baseline, Month 1, Month 2, Month 3, Month 4, Month 5, Month 6, Month 7, Month 8,Month 9, Month 10, Month 11, Month 12(end of treatment),Month 14(end of study),early termination visit (occurs only if subject discontinues form study)
  The SALT measures the percentage of hair loss on the scalp utilizing a visual aid showing the division of the scalp hair into four quadrants (back, top of scalp, and both sides), with each of the four quadrants given an accurate determination of the % of scalp surface area covered, representing 24%, 40%, 18%, and 18% of the total scalp surface area, respectively.
  Total SALT score is reported and calculated as: Total SALT Score=[0.40x%scalp hair loss top quadrant]+[0.24x%scalp hair loss back quadrant]+[0.18x%scalp hair loss left quadrant]+[0.18x% scalp hair loss right quadrant]
Number of subjects that achieved a 1-point increase in eyebrow assessment as assessed by the eyebrow assessment (EBA) score on the right side | Baseline, Month 1, Month 2, Month 3, Month 4, Month 5, Month 6, Month 7, Month 8,Month 9, Month 10, Month 11, Month 12(end of treatment),Month 14(end of study),early termination visit (occurs only if subject discontinues form study)
  This survey has a rating scale that ranges from 0 (none eyebrow) to 3 (normal eyebrow).This assessment will be performed for participants with eyebrows designated as one of the treatment areas, grading each eyebrow separately.
Number of subjects that achieved a 2-point increase in eyebrow assessment as assessed by the eyebrow assessment (EBA) score on the left side | Baseline, Month 1, Month 2, Month 3, Month 4, Month 5, Month 6, Month 7, Month 8,Month 9, Month 10, Month 11, Month 12(end of treatment),Month 14(end of study),early termination visit (occurs only if subject discontinues form study)
  This survey has a rating scale that ranges from 0 (none eyebrow) to 3 (normal eyebrow).This assessment will be performed for participants with eyebrows designated as one of the treatment areas, grading each eyebrow separately.
Number of participants with hair loss as described as a 1-point decrease in the Clinician Global Impression - Alopecia Areata (CGI-AA) | Baseline, Month 1, Month 2, Month 3, Month 4, Month 5, Month 6, Month 7, Month 8,Month 9, Month 10, Month 11, Month 12(end of treatment),Month 14(end of study),early termination visit (occurs only if subject discontinues form study)
  The Clinician Global Impression - Alopecia Areata (CGI-AA) is a single clinician-reported item developed to assess clinical impression of severity of scalp hair loss. The rater is asked to rate the participant's current hair loss on a 5 point static discrete scale ranging from 0 "None (no hair loss)", 1 "Minimal Hair Loss, 2 "Moderate Hair Loss", 3 "Severe Hair Loss" 4 "Very Severe or complete hair loss" with higher scores indicating more severe hair loss.
Number of participants with hair loss as described as a 2-point decrease in the Clinician Global Impression - Alopecia Areata (CGI-AA) | Baseline, Month 1, Month 2, Month 3, Month 4, Month 5, Month 6, Month 7, Month 8,Month 9, Month 10, Month 11, Month 12(end of treatment),Month 14(end of study),early termination visit (occurs only if subject discontinues form study)
  The Clinician Global Impression - Alopecia Areata (CGI-AA) is a single clinician-reported item developed to assess clinical impression of severity of scalp hair loss. The rater is asked to rate the participant's current hair loss on a 5 point static discrete scale ranging from 0 "None (no hair loss)", 1 "Minimal Hair Loss, 2 "Moderate Hair Loss", 3 "Severe Hair Loss" 4 "Very Severe or complete hair loss" with higher scores indicating more severe hair loss.

SECONDARY OUTCOMES:
AA as assessed by the Patient's Global Impression of Change (PGI-C) scale | Month 1, Month 2, Month 3, Month 4, Month 5, Month 6, Month 7, Month 8,Month 9, Month 10, Month 11, Month 12(end of treatment),Month 14(end of study),early termination visit (occurs only if subject discontinues form study)
  The Patient's Global Impression of Change (PGI-C) asks the participant to evaluate the improvement or worsening of their AA as compared to the start of the study using a single-item, "Since the start of the study, my alopecia areata has: …". The participants will select one of seven responses ranging from "greatly improved" to "greatly worsened."
Number of subjects with moderately improved AA as assessed by the Patient's Global Impression of Change (PGI-C) scale | Month 1, Month 2, Month 3, Month 4, Month 5, Month 6, Month 7, Month 8,Month 9, Month 10, Month 11, Month 12(end of treatment),Month 14(end of study),early termination visit (occurs only if subject discontinues form study)
  The Patient's Global Impression of Change (PGI-C) asks the participant to evaluate the improvement or worsening of their AA as compared to the start of the study using a single-item, "Since the start of the study, my alopecia areata has: …". The participants will select one of seven responses ranging from "greatly improved" to "greatly worsened."
Number of subjects with greatly improved AA as assessed by the Patient's Global Impression of Change (PGI-C) scale | Month 1, Month 2, Month 3, Month 4, Month 5, Month 6, Month 7, Month 8,Month 9, Month 10, Month 11, Month 12(end of treatment),Month 14(end of study),early termination visit (occurs only if subject discontinues form study)
  The Patient's Global Impression of Change (PGI-C) asks the participant to evaluate the improvement or worsening of their AA as compared to the start of the study using a single-item, "Since the start of the study, my alopecia areata has: …". The participants will select one of seven responses ranging from "greatly improved" to "greatly worsened."
Quality of life as assessed by the Dermatology Life Quality Index( DLQI) | Baseline,Mont4, Month 6, Month 9,Month 12
  The DLQI is a self administered validated questionnaire designed to measure the health-related quality of life of adult patients (greater than 16 years of age)suffering from a skin disease. This survey has 10 questions and each is scored on a 4 point scale from 0(not at all)-3(very much) for a maximum score of 30 and higher scores mean greater impairment of patient's quality of life
Quality of life as assessed by the Children's Dermatology Life Quality Index (CDLQI) | Baseline,Mont4, Month 6, Month 9,Month 12
  CDLQI is designed to measure the impact of any skin disease on the lives of children.This survey has 10 questions and each is scored on a 4 point scale from 0(not at all)-3(very much) for a maximum score of 30 and higher scores mean greater impairment of patient's quality of life
Quality of life as assessed by the Alopecia Areata Quality of Life Index (AA-QLI) | Baseline,Mont4, Month 6, Month 9,Month 12
  This is a 21 item questionnaire asking about whether they have a negative effect from alopecia scored categorically as very much, a lot, a little and not at all.Not at all indicating better quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Adelaide Hebert, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No